CLINICAL TRIAL: NCT00637858
Title: Effect of Different Doses of Tomato Lycopene on the Blood Pressure in Prehypertensives and Grade I Never Treated Otherwise Healthy Subjects
Brief Title: Effect of Different Doses of Tomato Lycopene on Blood Pressure in Pre-hypertensive Otherwise Healthy Subjects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty to enroll more subjects
Sponsor: Soroka University Medical Center (Other)
Collaborators: LycoRed Ltd. (Industry); The S. Daniel Abraham International Center for Health and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOR459407CTIL
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2009-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Lycopene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Placebo Comparator)
  Interventions: Other: Placebo
- 2 (Active Comparator): Lyc-o-Mato 5mg
  Interventions: Dietary Supplement: Lyc-O-Mato 5mg
- 3 (Active Comparator): Lyc-o-Mato 15mg
  Interventions: Dietary Supplement: Lyc-O-Mato 15mg
- 4 (Active Comparator): Lyc-o-Mato 30mg
  Interventions: Dietary Supplement: Lyc-O-Mato 30mg
- 5 (Active Comparator): Lycopene capsules (non Lyc-o-mato) 15 mg
  Interventions: Dietary Supplement: Lycopene capsules (non Lyc-o-mato) 15 mg

INTERVENTIONS:
Dietary Supplement: Lyc-O-Mato 5mg — Daily Lyc-O-Mato 5mg with lunch for 8 weeks (After 4 weeks of placebo run in). Lyc-O-Mato 6%, Natural tomato Complex, is packed into soft gelatin capsule
  Arms: 2
Dietary Supplement: Lyc-O-Mato 15mg — Daily Lyc-O-Mato 15mg with lunch for 8 weeks (After 4 weeks of placebo run in). Lyc-O-Mato 6%, Natural tomato Complex, is packed into soft gelatin capsule
  Arms: 3
Dietary Supplement: Lyc-O-Mato 30mg — Daily Lyc-O-Mato 30mg with lunch for 8 weeks (After 4 weeks of placebo run in). Lyc-O-Mato 6%, Natural tomato Complex, is packed into soft gelatin capsule
  Arms: 4
Dietary Supplement: Lycopene capsules (non Lyc-o-mato) 15 mg — Daily Lycopene capsules (non Lyc-o-mato) 15 mg with lunch for 8 weeks (After 4 weeks of placebo run in).
  Arms: 5
Other: Placebo — Placebo capsules, identical looking to previous capsules for double-blind treatment period (8 weeks) and single blind run-in (4 weeks).
  Arms: 1

SUMMARY:
Effect of different doses of tomato extract (contain Lyc-o-Mato 6% Oleoresin which Contain: 5, 15 mg lycopene , in addition to Beta-carotene (0.15%), phytoene, and phytofluene (1%); and vitamin E (2%), phospholipids (15%), and phytosterols (0.6%) suspended in tomato oleoresin oil) compared with synthetic lycopene on blood pressure and plasma lycopene levels in never treated pre-hypertensive otherwise healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35-60,
* No antihypertensive treatment in the past or present,
* 135< SBP< 145 or 85<DBP<95,
* Informed consent signed,

Exclusion Criteria:

* Unwilling to participate in the study,
* Treated essential,
* secondary or complicated hypertension,
* SBP lower than 135 or higher than 145 mmHg,
* DBP lower than 85 or higher than 95 mmHg,
* Use of other medications (statins, NSAI ect..),
* Known allergy to tomato, carotenoids, or vitamin E,
* Diabetes Mellitus,
* Obesity BMI>32,
* Significant dyslipidemia,
* Patients with ischemic pain, S/P MI, PTCA or CABG, LVH or CHF,
* Smoker,
* Valvular heart disease,
* PVD,
* Cerebrovascular disease, s/p CVA, TIA,
* Any kind of kidney disease (creatinine>1.6),
* Chronic liver disease(elevated AST and ALT at least by 2 times of the normal range),
* Alcohol abuse,
* History of GI disease or surgery,
* History of malignancy in the past 5 years,
* History of autoimmune disease,
* Participation in other researches protocol

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Every 2 weeks (Overall 12 weeks )

SECONDARY OUTCOMES:
Serum lycopene levels | Week 0,Week 12
Serum Phytofluene levels | Week 0,Week 12
Serum 8 isoprostane levels | Week 0,Week 12
Serum nitrite-nitrate levels | Week 0,Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Ester Paran, Professor, Principal Investigator — Hypertension clinic of the Soroka University Hospital
Locations (1):
- Hypertension Unit, Beersheba, Israel

REFERENCES:
- [Background] Engelhard YN, Gazer B, Paran E. Natural antioxidants from tomato extract reduce blood pressure in patients with grade-1 hypertension: a double-blind, placebo-controlled pilot study. Am Heart J. 2006 Jan;151(1):100. doi: 10.1016/j.ahj.2005.05.008. PMID 16368299